CLINICAL TRIAL: NCT07151274
Title: Impact of Ehlers-Danlos Syndrome on Gynaecological Health: Focus on the Prevalence of Dysmenorrhoea
Brief Title: Impact of Ehlers-Danlos Syndrome on Gynaecological Health
Acronym: GYNESED
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0124/OB; 2025-A00962-47 (Other: ANSM)
Record Dates: First submitted 2025-08-21; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Ehlers-Danlos Syndrome (EDS)
Keywords: gynaecological disorder; dysmenorrhea; menorrhagia; dyspareunia; endometriosis
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Dysmenorrhea; Menorrhagia; Dyspareunia; Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: women with Ehlers-Danlos syndrome (EDS): Women with Ehlers-Danlos syndrome (EDS) of all types diagnosed by a healthcare professional
- Comparator group: Women not affected by Ehlers-Danlos syndrome (EDS): Women without Ehlers-Danlos syndrome (EDS) (control group) from a healthy volunteer base

SUMMARY:
Dysmenorrhea is a common problem in gynaecology, significantly impacting patients' quality of life. Ehlers-Danlos syndrome (EDS) is associated with joint hypermobility, tissue fragility and chronic pain. Some studies suggest an increased prevalence of gynaecological disorders, including dysmenorrhea, in patients with EDS. However, data remain limited and few studies have compared the intensity and characteristics of dysmenorrhea in women with EDS. There is also little data on the prevalence of other gynaecological conditions in women with EDS.

This study therefore aims to compare the severity of dysmenorrhea in patients with EDS and a control group in order to better characterise the gynaecological impact of EDS. It will also compare the prevalence of other gynaecological conditions between women with EDS and women without EDS.

DETAILED DESCRIPTION:
Patients with SED report a high prevalence of gynaecological disorders, including severe dysmenorrhoea, menorrhagia and dyspareunia. Chronic pelvic pain and pelvic floor disorders are also common, impacting quality of life and reproductive function. Menorrhagia is common and may be due to capillary fragility and altered uterine connective tissue. The use of contraceptive hormones is often considered to reduce menstrual symptoms, although their effectiveness varies. A multidisciplinary approach is recommended to tailor treatments to the specific needs of patients.

Epidemiological data on the prevalence of EDS and hypermobility spectrum disorder show an increase in diagnoses, highlighting the importance of better clinical recognition.

Primary dysmenorrhoea is generally linked to excessive production of prostaglandins, leading to uterine hypercontractility and transient myometrial ischaemia. In patients with EDS, several pathophysiological mechanisms could contribute to exacerbated menstrual pain:

* Collagen dysregulation: fragility of uterine connective tissues that can alter myometrial contractility.
* Frequent dysautonomia in SED: may alter uterine vascularisation and amplify pain.
* Nociceptive hypersensitivity: described in patients with SED, increasing pain perception. This project hypothesises that patients with EDS experience more severe and/or more frequent dysmenorrhoea than the general population due to the tissue and neurological alterations specific to this syndrome.

Thus, evidence of increased dysmenorrhoea severity in EDS patients could justify better pain management and gynaecological care for these patients.

Better recognition of gynaecological disorders in EDS could prevent late diagnoses and therapeutic uncertainty.

Better recognition of gynaecological disorders in EDS could help to avoid late diagnoses and therapeutic uncertainty.

The prospects for this research are to show that a significant difference could be observed and to explore the underlying mechanisms (dysautonomia, local inflammation, myometrial abnormalities) in greater depth. The benefits of specialised gynaecological care with the introduction of hormone therapy could also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or over.
* Willing to participate voluntarily in the study via an online questionnaire.
* Of childbearing age.
* Reporting a diagnosis of EDS (all types) or not having EDS (control group) and being part of a database of healthy volunteers.

Exclusion Criteria:

* Minors (< 18 years old).
* Menopausal women
* People who do not understand French well enough to complete the questionnaire.
* Uncertain diagnosis of EDS (exclusion of participants who suspect EDS but without medical confirmation).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women diagnosed with Ehlers-Danlos syndrome (EDS)
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the severity of dysmenorrhea by Numerical Pain Scale (NPS) | Day 1
  The main objective of this study is to compare the severity of dysmenorrhea in patients with Ehlers-Danlos syndrome (EDS), all types combined, and a control group of patients without connective tissue disease. This comparison will determine whether EDS is a risk factor for more severe dysmenorrhea. The primary endpoint will be measured using the numerical pain scale (NPS), which assesses pain intensity on a scale of 0 to 10. A score of 10 corresponds to the "maximum imaginable pain"

SECONDARY OUTCOMES:
Analysis of clinical factors associated with the severity of dysmenorrhea (Age) using Numerical Pain Scale (NPS) | Day1
  Examine the impact of age on the intensity of dysmenorrhea, measured by the numerical pain scale (NPS). The outcome measure will be the Numerical Pain Scale (NPS), which rates pain intensity on a scale of 0 to 10. A score of 10 corresponds to the "maximum imaginable pain."
Analysis of clinical factors associated with the severity of dysmenorrhea (Body Mass Index (BMI)) using Numerical Pain Scale (NPS) | Day1
  Examine the impact of BMI on the intensity of dysmenorrhea, measured by the numerical pain scale (NPS). The outcome measure will be the Numerical Pain Scale (NPS), which rates pain intensity on a scale of 0 to 10. A score of 10 corresponds to the "maximum imaginable pain."
Analysis of clinical factors associated with the severity of dysmenorrhea (age of onset of dysmenorrhea,) using Numerical Pain Scale (NPS) | Day1
  Examine the impact of age of onset of dysmenorrhea, on the intensity of dysmenorrhea, measured by the numerical pain scale (NPS). The outcome measure will be the Numerical Pain Scale (NPS), which rates pain intensity on a scale of 0 to 10. A score of 10 corresponds to the "maximum imaginable pain."
Analysis of clinical factors associated with the severity of dysmenorrhea (presence of associated menorrhagia) using Numerical Pain Scale (NPS) | Day1
  Examine the impact of presence of associated menorrhagia on the intensity of dysmenorrhea, measured by the numerical pain scale (NPS). The outcome measure will be the Numerical Pain Scale (NPS), which rates pain intensity on a scale of 0 to 10. A score of 10 corresponds to the "maximum imaginable pain.".
Analysis of clinical factors associated with the severity of dysmenorrhea (medical history) using Numerical Pain Scale (NPS) | Day1
  Examine the impact of medical history on the intensity of dysmenorrhea, measured by the numerical pain scale (NPS). The outcome measure will be the Numerical Pain Scale (NPS), which rates pain intensity on a scale of 0 to 10. A score of 10 corresponds to the "maximum imaginable pain."
Study of the prevalence of gynaecological conditions (menorrhagia) | Day 1
  Evaluate the frequency of occurrence of a menorrhagia
Study of the prevalence of gynaecological conditions (endometriosis) | Day 1
  Evaluate the frequency of occurrence of endometriosis
Study of the prevalence of gynaecological conditions (adenomyosis) | Day 1
  Evaluate the frequency of occurrence of a adenomyosis
Study of the prevalence of gynaecological conditions (PolyCystic ovary syndrome (PCOS)) | Day 1
  Evaluate the frequency of occurrence of PCOS
Study of the prevalence of gynaecological conditions (abnormal cervical smear) | Day 1
  Evaluate the frequency of occurrence of abnormal cervical smear

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.